CLINICAL TRIAL: NCT03131362
Title: REALizing and Improving Management of Stable COPD in China--A Multi-centre, Prospective, Observational Study to Realize the Current Situation of COPD Patients in China.
Brief Title: Realize the Current Situation of COPD Patients in China
Acronym: REAL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D2287R00114
Record Dates: First submitted 2017-03-20; First posted 2017-04-27 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Chronic Obstructive Pulmonary Disease COPD
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-centre, prospective, observational study to realize the current situation of COPD patients in China. About 5000 COPD patients will be enrolled from 50 participating sites around China and followed up for one year. During this study, patients will undergo clinical assessments and receive medical care as determined by their treating physician.

DETAILED DESCRIPTION:
This is a multi-centre, prospective, observational study. This study aims to observe the general situation in clinical practice, and the evolution and outcome of current usual care of COPD in China.This is an observational study. It will be carried out under routine clinical practice and the treatment will be determined by patients' treating physicians. Information about exposure to treatments as part of routine care will be collected (dose, frequency and duration).

A multi-stage, stratified and cluster sampling method will be used to select a nationally representative sample from the tertiary and secondary hospitals with respiratory department in six geographic regions around China as the study sites. Approximately 5000 patients with COPD will be enrolled from 50 selected study sites in order to recruit a nationally representative study population and followed up for one year.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients, more than 40 years old
* Clinically diagnosed as COPD (the patients are clinically diagnosed as COPD based on chronic cough, sputum, wheeze and a history of exposure to harmful factors, and confirmed by spirometry(FEV1/FVC<0.7, post-bronchodilator according to GOLD 2016)
* Sign (or their legally-acceptable representatives must sign) and date the informed consent form indicating that they understand the purpose of and procedure required for the study and are willing to participate in the study.

Exclusion Criteria:

* Participated in any interventional clinical trial during the last 30 days
* With acute exacerbation within 4 weeks before enrolment
* Not suitable for study observation judged by investigators.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 5000 patients with COPD will be enrolled from 50 tertiary and secondary hospitals in six geographic regions around China in order to recruit a nationally representative study population from 2017 Q2 to 2018 Q2.
Sampling Method: Probability Sample
Enrollment: 5020 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-08-06 (Actual)

PRIMARY OUTCOMES:
The mean rate of COPD exacerbations | within one year
  The mean rate of COPD exacerbations (acute exacerbation number per patient per year).
The proportion of hospitalized patients | within one year
  The proportion of hospitalized patients due to the COPD exacerbations within one year；
The distribution of different severity of COPD exacerbations | within one year
  The distribution will be measured by percentage of patient on each level of severity of COPD exacerbations (mild: requiring an increase in rescue medication≥ 3 puffs / day for at least 2 consecutive days; moderate: requiring systemic glucocorticosteroids and/or antibiotics; severe: hospitalization, emergency room visit or leading to death), the calculation will be based on non-missing data.
The mean reduction value of available FEV1 | within one year
  The mean reduction value of available FEV1 after one year from baseline
The mean change in CAT | within one year
  The mean change in CAT total scores after one year from baseline; COPD assessment test (CAT) total score will be derived by summing up the score of all items. Total Scores range 0-40.The COPD influence on patients: 1 stage (mild): 0-10 points; 2 stage (moderate): 11-20 points; 3 stage (severe):21-30 points; 4 stage (very severe):31-40 points.
The mean change in mMRC | within one year
  The mean change in mMRC results after one year from baseline. Modified Medical Research Council Questionnaire (mMRC) will be assessed according to the severity of breathlessness as below:
  Grade 0 I only get breathless with strenuous exercise
  Grade 1 I get short of breath when hurrying on the level or walking up a slight hill
  Grade 2 I walk slower than people of the same age on the level because of breathlessness, or I have to stop for breath when walking on my own pace on the level
  Grade 3 I stop for breath after walking about 100 meters or after a few minutes on the level
  Grade 4 I am too breathless to leave the house or I am breathless when dressing or undressing
The mean change in COPD-Q | within one year
  The mean change in COPD patients' cognition questionnaire (COPD-Q) total scores after one year from baseline. COPD knowledge Questionnaire (COPD-Q) total score will be derived by summing up the scores from 13 items evaluating patients knowledge and understanding to COPD including 8 forward items: 1point (true), 0 point (false or not sure); 5 reverse items: 1 point (false), 0 point (true or not sure). Then get the total scores.
The mean rate of COPD exacerbations by different severity of COPD patients by airway limitation / by A/B/C/D at baseline. | within one year
  The mean rate of COPD exacerbations (acute exacerbation number per patient per year) by different severity of COPD patients by airway limitation / by A/B/C/D at baseline according to GOLD 2016.
The proportion of hospitalized patients by different severity of COPD patients by airway limitation / by A/B/C/D at baseline | within one year
  The proportion of hospitalized patients due to the COPD exacerbations by different severity of COPD patients by airway limitation / by A/B/C/D at baseline within one year according to GOLD 2016.
The mean reduction value of available FEV1 by different severity of COPD by airway limitation / by A/B/C/D patients after one year from baseline | within one year
  The mean reduction value of available FEV1 by different severity of COPD by airway limitation / by A/B/C/D patients according to GOLD 2016 after one year from baseline

SECONDARY OUTCOMES:
The distribution of different severity of COPD patients | within one year
  The distribution will be measured by the percentage of patient on each level of severity of COPD patients by airway limitation / by A/B/C/D patients at baseline and after one year. The calculation will be based on non-missing data.
Distribution of stable COPD medications in mono in total population by drug class | within one year
  The distribution will be measured by the percentage of patient on each kind of stable COPD medications in mono in total population by drug class (ICS[inhaled corticosteroid], LABA[long-acting beta2-agonist], ICS/LABA[combination long-acting beta2-agonists plus corticosteroids in one inhaler], SABA[short-acting beta2-agonist], SAMA[short-acting muscarinic antagonist], SABA/SAMA [combination short-acting beta2-agonist plus anticholinergic], LAMA[long-acting muscarinic antagonist], methylxanthines, mucolytic, traditional Chinese medicine and others [antibiotics, systemic corticosteroids, vaccines, antioxidant agents, etc]) at baseline and after one year. The calculation will be based on non-missing data.
Distribution of stable COPD medications by drug class according to the severity by airway limitation / by A/B/C/D patients | within one year
  The distribution will be measured by the percentage of stable COPD medications by drug class (ICS[inhaled corticosteroid], LABA[long-acting beta2-agonist], ICS/LABA[combination long-acting beta2-agonists plus corticosteroids in one inhaler], SABA[short-acting beta2-agonist], SAMA[short-acting muscarinic antagonist], SABA/SAMA [combination short-acting beta2-agonist plus anticholinergic], LAMA[long-acting muscarinic antagonist], methylxanthines, mucolytic, traditional Chinese medicine and others [antibiotics, systemic corticosteroids, vaccines, antioxidant agents, etc]) according to the severity by airway limitation / by A/B/C/D patients at baseline and after one year. The calculation will be based on non-missing data.
Distribution of medications for COPD exacerbations by drug class including hospital prescribed and pharmacy bought | within one year
  The distribution will be measured by the percentage of patient on each kind of medications for COPD exacerbations by drug (short-acting bronchodilators, corticosteroids, antibiotics and others) including hospital prescribed and pharmacy bought. The calculation will be based on non-missing data.
Distribution of non-drug treatments | within one year
  The distribution will be measured by the percentage of patient on each kind of non-drug treatments (health education, smoking cessation, exercise of respiratory function and vaccine injection) during the study. The calculation will be based on non-missing data.
Patients drug compliance | within one year
  Patients drug compliance (actual drug taken days/actually prescribed days, and actual drug taken dosage/actually prescribed dosage)
Mean total direct COPD cost | within one year
  Mean total direct COPD cost of the whole year per patient including the stable COPD management cost (medications and non-drug treatments) and the COPD exacerbations cost.
Distribution of prescribed stable COPD medications by drug class at each usual visit. | within one year
  The distribution will be measured by the percentage of patient on each kind of prescribed stable COPD medications by drug class (ICS[inhaled corticosteroid], LABA[long-acting beta2-agonist], ICS/LABA[combination long-acting beta2-agonists plus corticosteroids in one inhaler], SABA[short-acting beta2-agonist], SAMA[short-acting muscarinic antagonist], SABA/SAMA [combination short-acting beta2-agonist plus anticholinergic], LAMA[long-acting muscarinic antagonist], methylxanthines, mucolytic, traditional Chinese medicine and others [antibiotics, systemic corticosteroids, vaccines, antioxidant agents, etc]) on each usual care visit. The calculation will be based on non-missing data.
Distribution of stable COPD dosage by drug class according to the severity by airway limitation / by A/B/C/D patients at baseline and after one year. | Within one year
  The distribution will be measured by the percentage of patient on each kind of stable COPD dosage by drug class according to the severity by airway limitation / by A/B/C/D patients at baseline and after one year. The calculation will be based on non-missing data.
Distribution of stable COPD frequency by drug class according to the severity by airway limitation / by A/B/C/D patients at baseline and after one year. | Within one year
  The distribution will be measured by the percentage of patient on each level of stable COPD frequency by drug class ( same as above) according to the severity by airway limitation / by A/B/C/D patients at baseline and after one year.
  The calculation will be based on non-missing data.
Patients visit compliance | Within one year
  Patients visit compliance (the mean usual care visit times per patient per year, and the dropout rate at each visit including V0, V1 and TC visits)
Distribution of stable COPD medications in combination in total population by drug class | Within one year
  The distribution will be measured by the percentage of patient on each kind of stable COPD medications in combination in total population by drug class (ICS[inhaled corticosteroid], LABA[long-acting beta2-agonist], ICS/LABA[combination long-acting beta2-agonists plus corticosteroids in one inhaler], SABA[short-acting beta2-agonist], SAMA[short-acting muscarinic antagonist], SABA/SAMA [combination short-acting beta2-agonist plus anticholinergic], LAMA[long-acting muscarinic antagonist], methylxanthines, mucolytic, traditional Chinese medicine and others [antibiotics, systemic corticosteroids, vaccines, antioxidant agents, etc]) at baseline and after one year. The calculation will be based on non-missing data.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Yang T, Cai B, Cao B, Kang J, Wen F, Chen Y, Jian W, Wang C. REALizing and improving management of stable COPD in China: results of a multicentre, prospective, observational study (REAL). Ther Adv Respir Dis. 2023 Jan-Dec;17:17534666231178692. doi: 10.1177/17534666231178692. PMID 37318116
- [Derived] Yang T, Cai B, Cao B, Kang J, Wen F, Chen Y, Jian W, Wang C. Exacerbation in patients with stable COPD in China: analysis of a prospective, 52-week, nationwide, observational cohort study (REAL). Ther Adv Respir Dis. 2023 Jan-Dec;17:17534666231167353. doi: 10.1177/17534666231167353. PMID 37073797
- [Derived] Yang T, Cai B, Cao B, Kang J, Wen F, Chen Y, Jian W, Wang C. Treatment patterns in patients with stable COPD in China: analysis of a prospective, 52-week, nationwide, observational cohort study (REAL). Ther Adv Respir Dis. 2023 Jan-Dec;17:17534666231158283. doi: 10.1177/17534666231158283. PMID 37013442
- [Derived] Yang T, Cai B, Cao B, Kang J, Wen F, Chen Y, Jian W, Shang H, Wang C. Severity distribution and treatment of chronic obstructive pulmonary disease in China: baseline results of an observational study. Respir Res. 2022 Apr 29;23(1):106. doi: 10.1186/s12931-022-02021-w. PMID 35488337
- [Derived] Yang T, Cai B, Cao B, Kang J, Wen F, Yao W, Zheng J, Ling X, Shang H, Wang C. REALizing and improving management of stable COPD in China: a multi-center, prospective, observational study to realize the current situation of COPD patients in China (REAL) - rationale, study design, and protocol. BMC Pulm Med. 2020 Jan 13;20(1):11. doi: 10.1186/s12890-019-1000-x. PMID 31931767
- See also: This is a CSR Synopsis. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D2287R00114&attachmentIdentifier=91a8e174-23ff-4097-b401-63dcf2af3550&fileName=D2287R00114-Study_report_synopsis.pdf&versionIdentifier=